CLINICAL TRIAL: NCT04839328
Title: A Phase Ⅲ Multicenter, Randomized, Double-blind, Placebo-controlled To Assess Efficacy and Safety Study of Hemay005 in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Phase Ⅲ Efficacy and Safety Study of Hemay005 in Subjects With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tianjin Hemay Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HM005PS3S01
Record Dates: First submitted 2021-04-01; First posted 2021-04-09 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Hemay005

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 60mg Hemay005 (Experimental): Patients with chronic plaque psoriasis will be treated BID for 16 weeks with 60mg Hemay005 in first phase. Then will be treated BID for 36-week extension followed with 60mg of Hemay005.
  Interventions: Drug: 60mg Hemay005
- Placebo (Placebo Comparator): Patients with chronic plaque psoriasis will be treated BID for 16 weeks with placebo in first phase. Then will be treated BID for 36-week extension followed with 60mg of Hemay005.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 60mg Hemay005 — Hemay005 is a small molecule PDE4 inhibitor.
  Other Names: Hemay005 tablet
  Arms: 60mg Hemay005
Drug: Placebo — Placebos are the same as drugs, but contain no Hemay005.
  Other Names: placebo tablet
  Arms: Placebo

SUMMARY:
Hemay005 is a novel phosphodiesterase type 4(PDE4) inhibitor being developed for the treatment of psoriasis. After single asending dose and mutiple asending dose in health subjects. phase 2 results suggest Hemay005 60 mg BID has a higher curative effect trend，and adverse reactions were mild, so we choose 60 mg BID as Hemay005 phase 3 dosage And the patients with moderate to severe plaque psoriasis will be randomized into 2 cohorts(60mg BID and placebo) approximately 306 subjects will be enrolled (204 in 60mg BID and 102 in placebo). This study includes an 16-week treatment Period, then a 36-week Treatment Period without placebo.

DETAILED DESCRIPTION:
Hemay005 is a novel phosphodiesterase type 4(PDE4) inhibitor being developed for the treatment of psoriasis. After single asending dose and mutiple asending dose in health subjects. phase 2 results suggest Hemay005 60 mg BID has a higher curative effect trend，and adverse reactions were mild, so we choose 60 mg BID as Hemay005 phase 3 dosage And the patients with moderate to severe plaque psoriasis will be randomized into 2 cohorts(60mg BID and placebo) approximately 306 subjects will be enrolled (204 in 60mg BID and 102 in placebo). This study includes an 16-week treatment Period, then a 36-week Treatment Period without placebo.

Primary Objectives:

To evaluate the effectiveness of Hemay005 tablets 60 mg twice daily (BID) compared with placebo in patients with moderate to severe chronic plaque psoriasis.

Secondary objective：

1. Evaluate other efficacy characteristics of Hemay005 tablets 60 mg BID compared with placebo in patients with moderate to severe chronic plaque psoriasis.
2. Evaluate the safety of Hemay005 tablets 60 mg BID in patients with moderate to severe chronic plaque psoriasis.
3. To evaluate the population pharmacokinetics (PPK) characteristics of Hemay005 tablets 60 mg BID in patients with moderate to severe chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of signing the informed consent, the age was more than or equal to 18 years old, regardless of gender；
2. Stable plaque psoriasis with a history of more than 6 months (from the time of randomization)；
3. Screening and baseline PSAI ≥12, sPGA≥3（Moderate to Severe）,affected body surface area BSA≥10%；
4. All subjects must agree and commit to the use of a reliable contraceptive regimen. Women of childbearing potential must undergo monthly pregnancy testing during the study and agree to use two of the following methods of contraception throughout the study and for 90 days after the last dose of study drug. Reliable contraceptive regimen: vasectomy, abstinence, the use of condoms, intrauterine contraceptives (IUD), (Oral administration, patch, ring, injection, implantation) Barrier methods (diaphragm with spermicide, condom with spermicide)；
5. The subjects voluntarily participated in the study and signed the informed consent .

Exclusion Criteria:

1. Forms of psoriasis other than chronic plaque-type; (i.e., erythrodermic and guttate psoriasis, palmar, plantar or nail disease) at screening;
2. Investigator diagnosed as drug-induced psoriasis (including but not limited to new onset or aggravation of psoriasis caused by beta blockers, calcium channel inhibitors or lithium preparations);
3. Skin diseases, chronic diarrhea, serious digestive system diseases (such as active gastric ulcer, gastrointestinal bleeding, etc.), or other autoimmune inflammatory diseases that may interfere with clinical evaluation, according to the investigator;
4. The screening period was accompanied with active infection (such as bacterial infection, viral infection, fungal infection, etc., which required oral or intravenous treatment), and the investigator assessed that participation in this study may increase the risk of subjects;
5. Subjects with a history of tuberculosis or active tuberculosis (there were signs or symptoms of active tuberculosis judged by the researcher at the time of screening);
6. Use of prohibited treatments of this study;
7. History of congenital or acquired immunodeficiency;
8. Subjects couldn't limit their uv exposure during the study period ;
9. History of apremilast or Hemay005 tablets;
10. Subjects with conditions that may affect oral drug absorption, such as subtotal gastrectomy, clinically significant diabetic gastroenteropathy, or certain types of weight-loss surgery, such as gastric bypass surgery, do not include surgery that simply separates the stomach into separate Chambers, such as gastric banding surgery;
11. Subjects with tumor or history of malignancy (solid organ tumor or hematological tumor including myelodysplastic syndrome) in the past 5 years;
12. History of alcohol or drug abuse or dependence in the past year;
13. Subjects with a history of mental illness, suicidal behavior (including positive attempt, interrupted attempt or attempted suicide) or suicidal thoughts in the past 6 months were not suitable for clinical trials after the evaluation of the investigator; subjects with severe anxiety or depression during the screening period were assessed as severe anxiety or depression;
14. There are clinically serious, progressive or uncontrollable diseases in the screening period, including but not limited to respiratory system, cardiovascular system, endocrine system, blood system, musculoskeletal system and nervous system. According to the assessment of investigator, participating in this study may increase the risk of subjects or interfere with data interpretation;
15. In the screening period, human immunodeficiency virus (HIV) serological positive (i.e., HIV antibody positive);Evidence of hepatitis B virus infection: hepatitis B surface antigen (HBsAg) positive, or hepatitis B core antibody (HBcAb) positive and HBV-DNA above the upper limit of the normal range, or hepatitis B E antibody (HBeAb) positive and HBV-DNA above the upper limit of the normal range;Evidence of hepatitis C virus (HCV) infection: HCV antibody positive;
16. During the screening period, there were any of the following laboratory abnormalities:

    1. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2 times the upper limit of normal value, or total bilirubin > 1.5 times the upper limit of normal value;
    2. Serum creatinine > 1.2 times the upper limit of normal value;
    3. The hemoglobin of male patients was less than 8.5 g / dl (85.0 g / L), and that of female patients was less than 8.0 g / dl (80.0 g / L);
    4. WBC count < 3.0 × 109 / L or ≥ 14 × 109 / L;
    5. Platelet count < 100 × 109 / L
17. Female who were pregnant during lactation or pregnancy, or during the planned study period, or subjects who had sperm / egg donation plans during the study period;
18. Know allergic to active ingredient or excipient of the investigational product;
19. Participated in any other interventional clinical trial within 4 weeks or 5 pharmacokinetic / pharmacodynamic half lives before randomization (whichever is longer);
20. The investigator considered that there are any other conditions that are not suitable for participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who have 75% or more reduction in [Psoriasis area-and-severity index score (PASI)] (PASI75). | week 16
  The proportion of subjects who have a reduction of 75% or more from baseline in the psoriasis area-and-severity index score (PASI 75) at week 16.

SECONDARY OUTCOMES:
Proportion of subjects achieving an overall sPGA score of clear (0) or almost clear (1) with at least a 2-point reduction from baseline. | week 16
  The static Physician's Global Assessment (sPGA) rated the investigator's overall clinical assessment of a participants plaque thickness, erythema, and scaling on a 6-point scale ranging from 0 (clear, except for residual discoloration) to 5 (majority of plaques have severe thickness, erythema, and scale). To assign a sPGA score, the investigator examined all psoriatic lesions and assigned a severity score ranging from 0 to 5 for thickness, erythema, and scaling. Scores for thickness, erythema, and scaling are summed and the mean of these 3 scores equals the overall sPGA score. Decreases in sPGA correspond to clinical improvement.
Proportion of subjects who have 75% or more reduction in [Psoriasis area-and-severity index score (PASI)] (PASI75). | 1 year
  PASI-75 was defined as a ≥75% decrease in the PASI at visit from the baseline PASI and was calculated as: ([baseline PASI - visit PASI]/ baseline PASI) ×100%.
Proportion of subjects achieving an overall sPGA score of clear (0) or almost clear (1) with at least a 2-point reduction from baseline. | 1 year
  The SPGA score can determine the overall damage of psoriasis at a given time point，and higher SPGA scores mean a worse outcome.
Proportion of subjects who have 90% or more reduction in [Psoriasis area-and-severity index score (PASI)] (PASI90). | 1 year
  The PASI-90 was defined as a ≥90% decrease from baseline in the PASI score at the visit，and higher PASI scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: jianzhong Zhang, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No